CLINICAL TRIAL: NCT06692244
Title: Efficacy and Safety of Additive Manufacturing Personalized Titanium Mesh in Guided Bone Regeneration: a Randomized, Single-blind, Positive-controlled Prospective Study
Brief Title: Efficacy and Safety of Additive Manufacturing Personalized Titanium Mesh in Guided Bone Regeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital of Stomatology, Sun Yat-Sen University (Other)
Collaborators: Southern Medical University, China (Other); Meizhou People's Hospital (Other); Shenzhen Stomatology Hospital (Unknown); Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Wang Jinming, Chief Physician, Hospital of Stomatology, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GHKQ-202408-L3
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Alveolar Bone Atrophy; Guided Bone Regeneration
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized Titanium Mesh (Experimental): Preoperative CBCT datas of participants are obtained to design and manufacture personalized titanium meshes.Use additive-manufactured personalized titanium meshes for guided bone regeneration.
  Interventions: Procedure: Guided Bone Regeneration Surgery Using Additive-Manufactured Personalized Titanium Mesh
- Prefabricated Titanium Mesh (Active Comparator): Use prefabricated titanium mesh for guided bone regeneration.
  Interventions: Procedure: Guided Bone Regeneration Surgery Using Prefabricated Titanium Mesh

INTERVENTIONS:
Procedure: Guided Bone Regeneration Surgery Using Additive-Manufactured Personalized Titanium Mesh — Preoperative CBCT datas of participants are obtained to design and manufacture personalized titanium meshes.Use additive-manufactured personalized titanium meshes for guided bone regeneration.In the bone grafting surgery, the additive-manufactured personalized titanium mesh is used to secure the bone substitutes, with fixation screws used to secure the titanium mesh.
  Arms: Personalized Titanium Mesh
Procedure: Guided Bone Regeneration Surgery Using Prefabricated Titanium Mesh — In bone grafting surgery, prefabricated titanium mesh is used to fix the bone substitutes, and fixation screws are used to secure the titanium mesh.
  Arms: Prefabricated Titanium Mesh

SUMMARY:
This goal of this single-blind, simple randomized, positive-controlled prospective study is to evaluate the effects of additive-manufactured personalized titanium mesh and traditional titanium mesh in guided bone regeneration for large alveolar bone defects. The study will assess the short-term and long-term efficacy, safety, and incidence of complications of the additive-manufactured personalized titanium mesh, along with an analysis of risk factors. Participants will be followed up for two years after surgery with free-of-charge clinical and radiographic examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients missing single or multiple teeth with moderate to severe bone defects in the edentulous area requiring complex guided bone regeneration. （Moderate bone defects: bone loss with residual alveolar ridge width between 1 mm and 3 mm; severe bone defects: bone loss with residual alveolar ridge width ≤ 1 mm.）
2. The edge of the edentulous area within 1 mm is alveolar bone, with no adjacent tooth roots or nerve canals, ensuring complete retention of the personalized titanium mesh edge. The apical edge of the edentulous area within 2 mm is alveolar bone, with no nerve canals, ensuring that retention screws for the personalized titanium mesh can be designed in this area.
3. The patient and/or his/her guardian agrees to participate in this trial and signs the informed consent form.

Exclusion Criteria:

1. Patients with edentulism.
2. Patients with mild bone defects (residual alveolar ridge width greater than 3 mm).
3. Presence of acute or chronic infection in the surgical area.
4. Presence of acute or chronic infection in the teeth adjacent to the edentulous area.
5. Participation in similar trials or other interventional clinical trials within 30 days prior to signing the informed consent form.
6. History of metal allergies, severe allergy history, or severe immune deficiency.
7. Uncontrolled metabolic diseases, such as Type 1 diabetes or Type 2 diabetes (HbA1c ≥ 7% or fasting blood glucose ≥ 7 mmol/L despite medication control), severe liver or kidney dysfunction (ALT, AST > 2 times the upper limit of normal, serum creatinine above the upper limit of normal).
8. Long-term use of steroid medications.
9. History of drug abuse or alcoholism.
10. Pregnant or breastfeeding women.
11. Poor compliance.
12. Other conditions deemed unsuitable for participation by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Osteogenesis efficiency | 6 months after surgery
  Based on the oral CBCT imaging data, bone volume is reconstructed for preoperative, the day of surgery, and six months after surgery. Bone volume changes are assessed by using mimics as the bone resorption rate. The bone formation effectiveness is evaluated based on the bone resorption rate.

SECONDARY OUTCOMES:
Incidence of titanium mesh exposure | 14 days, 1 month, 6 months, 1 year, and 2 years after surgery
  Record and observe the exposure of the titanium mesh during the healing process.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Wang, Principal Investigator — Hospital of Stomatology, Sun Yat-Sen University
Locations (1):
- Hospital of Stomatology, Sun Yat-Sen University, Guangzhou, Guangdong, China